CLINICAL TRIAL: NCT03177928
Title: Functional and Morphological Cardiac Changes in Myeloproliferative Neoplasms
Brief Title: Cardiac Changes in Myeloproliferative Neoplasms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AKAli, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CCMPNS
Record Dates: First submitted 2017-05-25; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- study group (Active Comparator): patients with myeloproliferative neoplasms and reveal cardiac complications by using echocardiogram, intervention by using transthorathic echocardiography for all patients.
  Interventions: Device: Transthorathic echocardiogram
- control group (Active Comparator): patients with hematological disorders including myeloproliferative neoplasms without cardiac affection by using echocardiogram. Intervention will be in the form of using transthorath echocardiography with all patients to reveal any cardiac abnormalities.
  Interventions: Device: Transthorathic echocardiogram
- control group 2 (Active Comparator): healthy people from the same age and sex will be investigated using echocardiogram. Intervention will be in the form of using transthorathic echocardiography.
  Interventions: Device: Transthorathic echocardiogram

INTERVENTIONS:
Device: Transthorathic echocardiogram — In echocardiography lab and using transthoracic echocardiogram to reveal any cardiac changes in patients.

SUMMARY:
Myeloproliferative neoplasms are heterogeneous group of clonal hematopoietic stem cell neoplasms with excessive proliferation of one or more of the erythroid, megakaryocytic, or myeloid lineages and relatively normal maturation resulting in increased numbers of red cells, platelets, and/or granulocytes in the peripheral blood. Constitutive tyrosine kinase activation appears to be a common pathogenetic mechanism.

DETAILED DESCRIPTION:
According to worldwide study of prevalence of myeloproliferative neoplasms revealed:

Incidence of polycythemia vera ranged 0.01 to 2.61 per 100.000 population and the prevalence ranging from 0.49 to 46.88 per 100.000 population. Incidence of essential thrombocythemia is 0.21 to 2.27 per 100.000 population, prevalence ranging between 11.00 - 42.51 per 100.000 population.

Primary myelofibrosis incidence is 1.15 -4.99 per 100.000 population and prevalence ranging between 1.76 - 4.05 per 100.000 population.In previous studies, cardiac involvement including coronary arterial thrombosis, myocardial infarction, pulmonary hypertension, asymptomatic pericardial effusion, cardiac tamponade, intractable cardiac failure due to intraventricular stenosis and valvular stenosis that occur in myeloproliferative neoplasms. There is a few number of studies in which cardiac lesions were evaluated in myeloproliferative neoplasms by using transthoracic echocardiography but still inadequate, so we need to understand more about cardiovascular complications in myeloproliferative neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria of myeloproliferative neoplasms.

Exclusion Criteria:

* Extreme body weight e.g., morbid obesity.
* Cardiac disease.
* Cerebrovascular disorders.
* Diabetes mellitus.
* Dyslipidemia.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-08-31 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
number of patients with cardiac complications in myeloproliferative diseases. | 30 minutes
  cardiac complications as valvular changes, ejection fraction changes, pulmonary hypertension

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] How common are myeloproliferative neoplasms? A systematic review and meta-analysis. Am J Hematol. 2015 Sep;90(9):850. doi: 10.1002/ajh.23984. Epub 2015 Mar 30. No abstract available. PMID 26299877
- [Background] Passamonti F, Maffioli M. Update from the latest WHO classification of MPNs: a user's manual. Hematology Am Soc Hematol Educ Program. 2016 Dec 2;2016(1):534-542. doi: 10.1182/asheducation-2016.1.534. PMID 27913526
- [Background] Campbell A. Now I know why. Front Nurs Serv Q Bull. 1968 Winter;43(3):7-9. No abstract available. PMID 5183970
- [Background] Titmarsh GJ, Duncombe AS, McMullin MF, O'Rorke M, Mesa R, De Vocht F, Horan S, Fritschi L, Clarke M, Anderson LA. How common are myeloproliferative neoplasms? A systematic review and meta-analysis. Am J Hematol. 2014 Jun;89(6):581-7. doi: 10.1002/ajh.23690. PMID 24971434
- [Background] Mehta J, Wang H, Iqbal SU, Mesa R. Epidemiology of myeloproliferative neoplasms in the United States. Leuk Lymphoma. 2014 Mar;55(3):595-600. doi: 10.3109/10428194.2013.813500. Epub 2013 Jul 29. PMID 23768070
- [Background] Barbui T, Thiele J, Gisslinger H, Finazzi G, Vannucchi AM, Tefferi A. The 2016 revision of WHO classification of myeloproliferative neoplasms: Clinical and molecular advances. Blood Rev. 2016 Nov;30(6):453-459. doi: 10.1016/j.blre.2016.06.001. Epub 2016 Jun 11. PMID 27341755